CLINICAL TRIAL: NCT02225548
Title: An Open-label Trial of Oral Selegiline 5 or 10 mg and Tadalafil 2.5mg Co-administration to Male Patients With Parkinson's Disease and Moderate Erectile Dysfunction.
Brief Title: Sagene 2014 - Parkinson's Disease and Erectile Dysfunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sagene 2014
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Parkinson's Disease; Erectile Dysfunction
MeSH Terms: conditions — Parkinson Disease; Erectile Dysfunction | interventions — Selegiline; Tadalafil

ARMS (1):
- Selegiline and Tadalafil (Experimental): Tadalafil 2.5mg for 4 weeks then oral selegiline 5mg daily for 2 weeks then increased to 5mg twice daily for 2 more weeks
  Interventions: Drug: Selegiline; Drug: Tadalafil

INTERVENTIONS:
Drug: Selegiline
  Other Names: Eldepryl; Zelapar
Drug: Tadalafil
  Other Names: Cialis; Adcirca

SUMMARY:
The purpose of this study is to see if selegiline and tadalafil (generic for Cialis®) results in an improvement in Erectile dysfunction (ED) in male patients with Parkinson's disease (PD) and moderate ED. Male PD patients who have an incomplete response to tadalafil alone will be given both medications to see if the addition of selegiline improves ED symptoms more than tadalafil alone. It is common practice for a medical doctor to prescribe these two drugs to a patient like you. However, there have been no studies conducted to examine the effects of these medications when taken together.

Selegiline is normally prescribed for PD patients that are taking carbidopa/levodopa who are not receiving complete benefit from carbidopa/levodopa.

Tadalafil is normally prescribed to men who have erectile dysfunction and/or benign prostatic hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of idiopathic Parkinson's disease that is optimally treated (motor fluctuations <20% of subject's awake time). Subjects may be on levodopa therapy but must be stable at the time of entry into the study
* Sexually active (i.e. ≥1 attempt/week) males, 40 - 64 years of age (inclusive) at time of screening
* Diagnosis of moderate erectile dysfunction (defined according to the NIH Consensus Development Panel on Impotence) for more than 6 months and demonstrating and incomplete response to tadalafil alone
* Subject demonstrating an IIEF-5 drug-free baseline score that is ≥ 10 but ≤ 16, and an IIEF-5 tadalafil-alone baseline score that is ≤ 18
* Subject in a stable heterosexual relationship for at least 6 months. (2)
* Subject motivated to seek treatment for erectile dysfunction.
* Subject with a total serum testosterone level ≥ 300 ng/dL, with or without supplementation
* Hoehn and Yahr Scale score of 1 - 3
* Patient able to consent and comply with protocol requirements

Exclusion Criteria:

* Subject unwilling to cease use of any treatment for erectile dysfunction during the study, including oral medication, vacuum devices, constrictive devices, injections, urethral suppositories, gels, any over-the-counter or nonprescription medications, and products purchased via the internet
* Subject receiving dopamine agonists, nitrates, alpha-receptor blocking agents, or antihypertensive medication (see other exclusionary medications listed below)
* Subject with a history of syncope within the last 6 months prior to screening
* Subject with symptomatic postural hypotension (severe dizziness or fainting
* Subject with hypotension and a resting systolic blood pressure of < 90 mmHG or hypertension with a resting systolic blood pressure > 170 mmHG or a resting diastolic blood pressure > 110 mmHG
* Subject with any underlying cardiovascular condition, including unstable angina pectoris, which preclude sexual activity
* Subject with a history of myocardial infarction, stroke or life-threatening arrhythmia within 6 months prior to screening
* Subject with uncontrolled atrial fibrillation/flutter at screening (defined as ventricular response rate ≥ 100 bpm)
* Subject with a bleeding disorder
* Subject with a history of prostatectomy because of prostate cancer, including nerve sparing techniques. Subjects with a history of surgical procedures for the treatment of benign prostate hypertrophy are permitted, with the exception of cryosurgery, cryotherapy or cryoablation
* Subject with hereditary degenerative retinal disorders such as retinitis pigmentosa
* Subject with a history of loss of vision because of non-arteritic anterior ischemic optic neuropathy (NAION), history of temporary or permanent loss of vision, including unilateral loss of vision
* Subject with a history of congenital QT prolongation
* Subject with a penile anatomical abnormality (e.g., penile fibrosis, fractures, or Peyronie's disease) which, in the investigator's opinion, could significantly impair sexual performance. This will be based on subject's reported medical history (penile exam not required)
* Subject with primary hypoactive sexual desire.
* Subject with a spinal cord injury
* Subject with a severe chronic or acute liver disease, history of moderate (Child-Pugh B), or severe (Child-Pugh C) hepatic impairment
* Subject with clinically significant chronic hematological disease which could lead to priapism such as sickle cell anemia, multiple myeloma, and leukemia
* Subject with active peptic ulceration
* Subject with a history of malignancy within the past 5 years (other than squamous or basal cell skin cancer)
* Subject with a history of a positive test for Hepatitis B surface antigen (HbsAg) or Hepatitis C
* Subject with a known hypersensitivity to any component of the investigational medications, monoamine oxidase inhibitors, phosphodiesterase type 5 inhibitors or phenylethylamines
* Subjects with a history of drug or alcohol abuse within the past 6 months
* Subjects currently consuming ≥5 units of alcohol per day
* Subject who is illiterate or unable to understand the Informed Consent Form, questionnaires or subject diary
* Subject who, in the opinion of the investigator, will be noncompliant with the visit schedule or study procedures
* Subject with any unstable medical, psychiatric, or substance abuse disorder that in the opinion of the investigator is likely to affect the subject's ability to complete the study or preclude the subject's participation in the study
* Diagnosis of any other neurologic disease
* Uncontrolled Diabetes (Hemoglobin A1C > 7.5)

Ages: 40 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Changes in International Index of Erectile Function-5 (IIEF-5) score between baseline (Week 8) to end-of-study (Week 16). | The IIEF-5 will be administered at Weeks 4, 8, 12 and 16 of the study.
  The International Index of Erectile Function (IIEF) is a widely used, multi-dimensional self-report instrument for the evaluation of male sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Zesiewicz, MD, FAAN, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States